CLINICAL TRIAL: NCT02917239
Title: Prevalence Analysis of Ocular Disorders in Patients on Treatment for Symptomatic Multiple Myeloma
Brief Title: Prevalence of Ocular Disorders in Multiple Myeloma (MM-OO-16)
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Vittorio Montefusco, Medical Doctor, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: MM-OO-16
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Overall survival of multiple myeloma (MM) patients has increased significantly due to the availability of the new drugs. Moreover, since MM is an incurable disease, patients are exposed to repeated lines of therapy with different agents. It is therefore increasingly important to monitor the long-term side-effects of treatments. In the present study we focused on ocular disorders. This is an observational study aiming to assess the prevalence of ocular disorders in 100 patients on treatment or follow-up for MM.

DETAILED DESCRIPTION:
This is an observational study aiming to assess the prevalence of ocular disorders in patients on treatment or follow-up for MM.

Study population Patients diagnosed with multiple myeloma on treatment and/or on follow-up after treatment for multiple myeloma. The study aims to enroll 100 patients.

Endpoints Primary endpoint: To determinate prevalence and main characteristics of ocular disorders in patients on treatment / or previously treated for Multiple Myeloma.

Secondary endpoints:

1. To evaluate the relation between the kind of treatment for multiple myeloma and the development of ocular disorders
2. To evaluate the relation between patient's characteristics and comorbidities (such as sex, age, smoking, hypertension, diabetes, autoimmune diseases) and the presence of ocular disorders in this population of patients.

Study design Patients will be enrolled in the study at any time starting for the 3rd month of treatment, regardless if they are still on treatment or not.

Patients will undergo an ocular evaluation including visual acuity analysis, evaluation of the anterior ocular segment, fundus oculi analysis, ocular pressure measurement, Schirmer's Test.

If clinically required by the ophthalmologist, the patient will also undergo:

* Optical computerized tomography
* Fundus autofluorescence
* Fluorescein angiography
* Computerized visual field

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of Multiple Myeloma
* Patients have started an active treatment for Multiple Myeloma since at least two months
* Patients on active treatment for relapsed/refractory multiple myeloma
* Patients on follow-up after previous active treatment for multiple myeloma

Exclusion Criteria:

* Bilateral blindness preceding the diagnosis of multiple myeloma
* No signature of the informed consent
* Patients have started an active treatment for Multiple Myeloma since less than two months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with symptomatic multiple myeloma on treatment and/or on follow-up after treatment for multiple myeloma.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To assess prevalence of reduced visual acuity (>/= 20/40), cataract (graded according to LOCS III grading scale), dry eye, retinopathy, elevated intraocular pressure (> 21 mmHg) in patients on treatment for Multiple Myeloma | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Montefusco, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano

IPD SHARING:
Plan to Share IPD: No